CLINICAL TRIAL: NCT05596071
Title: Whether Opioids Are Factor That Induced Postoperative Delirium?
Brief Title: Whether Opioids Are Factor That Induced POD?
Acronym: POD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Fang Jun, Director, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2016-10-10
Record Dates: First submitted 2021-06-22; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Delirium
Keywords: opioid; POD; gastric cancer
MeSH Terms: conditions — Emergence Delirium; Stomach Neoplasms | interventions — Sufentanil; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sufentanyl+Epidural analgesia (Experimental): Combined use of sufentanil and ropivacaine for intraoperative and postoperative analgesia
  Interventions: Drug: Sufentanil Citrate; Drug: Ropivacaine 0.75% Injectable Solution; Procedure: Epidural catheter
- Epidural analgesia (Sham Comparator): Only use of ropivacaine for intraoperative and postoperative analgesia
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution; Procedure: Epidural catheter

INTERVENTIONS:
Drug: Sufentanil Citrate — Intraoperative loading dose of sufentanil 0.6μg/kg, each additional hour 10μg, within one hour of the end of surgery to stop additional.Postoperative analgesia pump formula: sufentanil 150ug + 0.75% ropivacaine 60ml with 0.9% saline diluted to 220ml, 3ml
  Other Names: Sufentanil
  Arms: Sufentanyl+Epidural analgesia
Drug: Ropivacaine 0.75% Injectable Solution — Intraoperative epidural analgesia was performed with 0.5% ropivacaine 5-20 ml,Postoperative analgesia pump formula:0.75% ropivacaine 60ml with 0.9% saline diluted to 220ml, 3ml/h, Blos 3ml, locking time 15min, the maximum dose of 36ml in 4 hours Saline is used to dilute other drugs
  Other Names: Ropivacaine
Procedure: Epidural catheter — Intraoperative and postoperative analgesia

SUMMARY:
The purpose of this study was to investigate whether perioperative use of low doses of opioids could reduce postoperative delirium .

DETAILED DESCRIPTION:
Postoperative delirium (POD) is a common postoperative complication of the elderly caused by a variety of factors. POD is an acute neuropsychiatric disorder characterized by disturbance of attention consciousness and cognitive function fluctuation, and more than 40% of elderly patients have symptoms of hypoactivity POD.The incidence of POD is as high as 17% to 61% in patients with neurocognitive impairment and patients undergoing complex or emergency surgery, which usually occurs between 1 and 3 days after surgery. POD will lead to prolonged hospital stay, functional impairment and even death. How to prevent and treat POD is an urgent clinical problem to be solved at present.

Opiates are commonly used perioperative sedatives and analgesics, which may be associated with the occurrence of postoperative POD in elderly patients and increase the risk of POD. It is not clear whether perioperative use of low doses of opioids could reduces the incidence of POD in elderly patients. In this study, reducing-opioids anesthesia was defined as the use of 1/3 of the conventional opioid dose to observe whether reducing-opioids anesthesia affected the incidence of POD in elderly patients undergoing gastric cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ≥65 years
* Underwent elective radical gastrectomy

Exclusion Criteria:

* Mini-Mental Scale Test (MMSE) Exclusion criteria: illiteracy <18, primary school <21, junior school and above <25
* Preoperative clear systems and spiritual history of neurological disease or long-term use of sedatives or antidepressants
* History of alcohol abuse or a history of drug dependence
* Have brain surgery or trauma
* Cannot with the completion of tests of Postoperative Cognitive Dysfunction
* Refused to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-06-25 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 3 days after surgery
  confusion assessment method for the ICU(CAM-ICU)
Incidence of postoperative delirium | 3 days after surgery
  Richmond agitation and sedation scale(RASS), the RASS score was divided into 10 sedation scales, ranging from +4 to -5, representing the patient's degree from "aggressive" to "unconscious," with each score corresponding to a state of consciousness. When the RASS score was ≥-3, the CAM-ICU assessment was performed.

SECONDARY OUTCOMES:
Visual analogue scale(VAS) | 3 days after surgery
  VAS is a scale of 11 numbers ranging from 0 to 10, with 0 representing no pain and 10 representing the most pain. Patients choose one of the 11 numbers to represent the pain level according to their own pain.
  0: no pain;
  Less than 3 points: mild pain, tolerable;
  4-6 points: the patient's pain and affect sleep, still tolerable;
  7-10: Patients have increasing pain, pain is unbearable, affect appetite, affect sleep.
Anaesthesia related adverse event | 3 days after surgery
  Nausea and vomiting
blood pressure | 3 days after surgery
  Hypertension or hypotension was defined as an increase or decrease in mean arterial pressure of more than 30% at baseline

CONTACTS AND LOCATIONS:
Overall Officials: chaoqun Fei, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
this study individual statistics is not available